CLINICAL TRIAL: NCT04535622
Title: A Randomized Controlled Trial to Evaluate Effect of a Structured Rehabilitation Exercise Program on Facedown Posture-related Pain After Retinal Surgery
Brief Title: Efficacy of Exercise Program for Facedown Posture-related Pain After Retinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Se Woong, Kang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-03-157
Record Dates: First submitted 2020-08-26; First posted 2020-09-02 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Macular Holes; Retinal Detachment
Keywords: face-down posture; musculoskeletal pain; vitrectomy
MeSH Terms: conditions — Retinal Perforations; Retinal Detachment; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the interventions participants and researchers cannot be blinded to group allocation. The treating healthcare professionals (i.e. the Research Nurse and Clinical Research Fellow) will also not be masked due to nature of the service. The surgeon will be masked to allocation. The data manager and trial statistician will be masked to allocation throughout the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): A structured exercise instruction for facedown posture-related pain will be provided to the patients, and patients will go through three times of self-exercise sessions everyday according to the training provided.
  Interventions: Behavioral: A structured exercise
- Control group (No Intervention): Patients are going to maintain face-down posture but no specific exercise instruction will be provided.

INTERVENTIONS:
Behavioral: A structured exercise — Exercise training will be conducted by a physical therapist which will take about 10 to 15 minutes. Patient education will include how to keep face down in various postures, and how to actively exercise the related muscles and joints while maintaining face-down posture through video clip and brochure. Patients will go through three times of self-exercise sessions everyday according to the training provided to the patients. Active exercise for the FDP patients will include exercise in a hands and knees position, limb exercise in an FDP, and exercise in a standing position. The exercises were performed within the range of individual muscle strength and fitness.
  Arms: Exercise group

SUMMARY:
The purpose of this study is to evaluate the effects of a structured exercise program on musculoskeletal pain of patients in face-down posture after retinal surgery.

DETAILED DESCRIPTION:
After being informed about the study, patients who are planning to get vitrectomy for macular hole or retinal detachment are going to be randomly assigned into two groups; exercise group and control group. All patients are going be admitted to the hospital prior to the surgery. After the surgery is done, the patients are going to maintain a face-down position in the ward until postoperative day 3. After returning to the ward after surgery and completed the pain scoring forms, exercise training is going to be conducted for patients assigned to the exercise group by a physical therapist. Three times of daily self-exercise sessions are going to be performed according to the training provided to the patients. Pain score will be measured on the first, second and the third postoperative days. Patients will be discharged on the third postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are getting vitrectomy for macular hole or retinal detachment and planning to maintain face-down posture.

Exclusion Criteria:

* Pre-existing musculoskeletal disorder.
* low visiual acuity in the opposite eye (best-corrected visual acuity less than 20/200 by snellen chart) making patients hard to get the exercise training.
* Patients with posture prescriptions other than the prone position

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Final pain score at back neck, shoulder, and lower back | postoperative day 3
  Pain score (numerical rating scale) at back neck, shoulder, and lower back at postoperative day 3 (discharge day). Possible scores range from 0 (no pain) to 10 (worst possible pain).

SECONDARY OUTCOMES:
pain score at back neck, shoulder, and lower back right on surgery day | surgery day
  Pain score based on numerical rating scale at back neck, shoulder, and lower back at postoperative day 1. Possible scores range from 0 (no pain) to 10 (worst possible pain).
pain score at back neck, shoulder, and lower back on postoperative day 1 | postoperative day 1
  Pain score based on numerical rating scale at back neck, shoulder, and lower back at postoperative day 2. Possible scores range from 0 (no pain) to 10 (worst possible pain).
pain score at back neck, shoulder, and lower back on postoperative day 2 | postoperative day 2
  Pain score based on numerical rating scale at back neck, shoulder, and lower back at postoperative day 2. Possible scores range from 0 (no pain) to 10 (worst possible pain).

OTHER OUTCOMES:
Patients satisfaction on the exercise program | postoperative day 3
  4 questionnaire items are as follow:
  1. The rehabilitation program help patients recover health. Answer: [1: strongly disagree 2: disagree 3: neither agree nor disagree 4: agree 5: strongly disagree]
  2. I want this exercise program the next time I have retinal surgery Answer: [1: strongly disagree 2: disagree 3: neither agree nor disagree 4: agree 5: strongly disagree]
  3. I would recommend this program to other patients getting retinal surgery Answer: [1: strongly disagree 2: disagree 3: neither agree nor disagree 4: agree 5: strongly disagree]
  4. Overall satisfaction Answer: [1: very disappointed 2: disappointed 3: neither satisfied nor disappointed 4: satisfied 5: very satisfied]

CONTACTS AND LOCATIONS:
Overall Officials: Se Woong Kang, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No